CLINICAL TRIAL: NCT01112969
Title: OSCAR - An Internet-based Supportive Coaching for Informal Caregivers of Adult Individuals With an Acquired Brain Injury.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Project end after 3 years; prolongation was rejected
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Prof. Dr. Hansjoerg Znoj, University of Bern, Department of Clinical Psychology and Psychotherapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSCAR; SNF-100014-124574, 2009-2012; 1784 -Bern University Hospital
Record Dates: First submitted 2010-04-05; First posted 2010-04-29 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Caregivers; Brain Injury
Keywords: Internet-based supportive coaching; guided self-help; Caregivers; Brain Injury; Caregiver Burden; Coping; Stress; Depression
MeSH Terms: conditions — Brain Injuries; Caregiver Burden; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based supportive coaching OSCAR (Experimental): Arm 1: Internet-based supportive coaching OSCAR
  Interventions: Behavioral: Internet-based supportive coaching OSCAR
- Waiting list control group (treatment as usual, TAU) (Other)
  Interventions: Other: Waiting-list control group (TAU)

INTERVENTIONS:
Behavioral: Internet-based supportive coaching OSCAR — The Internet-based supportive coaching (OSCAR) is an scientifically based multicomponent intervention
  Arms: Internet-based supportive coaching OSCAR
Other: Waiting-list control group (TAU) — Waiting-list control group (treatment as usual, TAU, no specific intervention)
  Arms: Waiting list control group (treatment as usual, TAU)

SUMMARY:
This is an intervention study for informal caregivers of adult patients with an acquired brain injury (stroke, traumatic brain injury or cerebral haemorrhage). It will determine whether an internet-based supportive coaching offers benefits to the caregivers in their own process of coping in the aftermath of a brain injury of a close relative. We expect the internet-based supportive coaching to be more effective in the treatment of emotional distress reactions and caregiver burden than the treatment as usual.

DETAILED DESCRIPTION:
Background

A brain injury (e.g. stroke, traumatic brain injury) occurs all of a sudden and is often followed by complex neurological and psychological consequences. These consequences do not only affect the patients with the brain injury as Muriel Lezak already stated in 1988: "Brain damage is a family affair". Symptoms of depression and anxiety as well as an increased caregiver burden are common, but there is still a lack in randomized controlled trials that investigate the efficacy of multicomponent interventions for informal caregivers. The main aim of the current study is to close this scientific gap with an innovative method for this special population. OSCAR (the Internet-based supportive coaching) uses the Internet as a communication- and information brokering medium and is designed as a "guided-self-help tool" where a qualified therapist individually supports every participant. The key objective is to investigate the feasibility, acceptance and efficacy of an Internet-based supportive coaching (OSCAR) for informal caregivers of adult individuals with an acquired brain injury. It is expected that the Internet-based supportive coaching (OSCAR) leads to a better coping of emotional distress reactions and caregiver burden.

Objective

A key objective is to investigate the feasibility, acceptance and efficacy of an Internet-based supportive coaching (OSCAR) for informal caregivers of adult individuals with an acquired brain injury.

Methods

To one part, OSCAR is part of a randomized controlled intervention study where a standard neuropsychological therapy is compared with an integrative neuro-psychotherapy. The Internet-based supportive coaching (OSCAR) for the caregivers is part of the integrative neuro-psychotherapy arm.

Additionally a randomized controlled intervention study with a waiting list-control-group design is realised.

Assessments will be made at baseline, after 4 months (progress), after ending with the training (termination) and at 6 months post treatment (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Family caregiver of an adult with a stroke, cerebral haemorrhage or traumatic brain injury
* sufficient German language skills
* at least 3 months after the brain injury
* access to a computer with internet access
* minimum age of 18 years
* informed consent to participate voluntarily in the study

Exclusion Criteria

* acute suicidal tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
German Zarit Burden Interview (G-ZBI) | Baseline
  The German Zarit Burden Interview (G-ZBI) is based on the Zarit Burden Interview (ZBI), the most widely used measure to assess caregiver burden. The 22 Items ask for the strain caregivers perceive (e.g., "Do you feel that your social life has suffered because you are caring for your relative?"). Responses range from 0 (never) to 4 (nearly always), the maximum score being 88. The higher the total score, the heavier the perceived burden.
German Zarit Burden Interview (G-ZBI) | 4 months after baseline
  The German Zarit Burden Interview (G-ZBI) is based on the Zarit Burden Interview (ZBI), the most widely used measure to assess caregiver burden. The 22 Items ask for the strain caregivers perceive (e.g., "Do you feel that your social life has suffered because you are caring for your relative?"). Responses range from 0 (never) to 4 (nearly always), the maximum score being 88. The higher the total score, the heavier the perceived burden.
German Zarit Burden Interview (G-ZBI) | 8 months after baseline
  The German Zarit Burden Interview (G-ZBI) is based on the Zarit Burden Interview (ZBI), the most widely used measure to assess caregiver burden. The 22 Items ask for the strain caregivers perceive (e.g., "Do you feel that your social life has suffered because you are caring for your relative?"). Responses range from 0 (never) to 4 (nearly always), the maximum score being 88. The higher the total score, the heavier the perceived burden.
German Zarit Burden Interview (G-ZBI) | 14 months after baseline (follow-up)
  The German Zarit Burden Interview (G-ZBI) is based on the Zarit Burden Interview (ZBI), the most widely used measure to assess caregiver burden. The 22 Items ask for the strain caregivers perceive (e.g., "Do you feel that your social life has suffered because you are caring for your relative?"). Responses range from 0 (never) to 4 (nearly always), the maximum score being 88. The higher the total score, the heavier the perceived burden.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) | Baseline
  The Beck Depression Inventory (BDI-II) is the 1996 revision of the BDI created by Dr. Aaron T. Beck, which is one of the most widely used self-report questionnaires measuring the severity of depression. The 21 multiple-choice items address the severity of 21 typical symptoms of depression over the past two weeks. The higher the total score, the more severe the depression.
Quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | Baseline
  The WHOQOL-BREF self-report questionnaire is the abbreviated 26-item version of the WHOQOL-100. It assesses the perceived quality of life (e.g. "To what extent do you feel your life to be meaningful?"). Quality of life is defined by the WHO as "…individuals' perceptions of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns."
Perceived Stress Questionnaire (PSQ20) | Baseline
  The Perceived Stress Questionnaire (PSQ20) is the abbreviated 20-item version of the PSQ (Levenstein et al., 1993) and assesses self-reported experienced stress.
Beck Depression Inventory (BDI-II) | 4 months after baseline
  The Beck Depression Inventory (BDI-II) is the 1996 revision of the BDI created by Dr. Aaron T. Beck, which is one of the most widely used self-report questionnaires measuring the severity of depression. The 21 multiple-choice items address the severity of 21 typical symptoms of depression over the past two weeks. The higher the total score, the more severe the depression.
Beck Depression Inventory (BDI-II) | 8 months after baseline
  The Beck Depression Inventory (BDI-II) is the 1996 revision of the BDI created by Dr. Aaron T. Beck, which is one of the most widely used self-report questionnaires measuring the severity of depression. The 21 multiple-choice items address the severity of 21 typical symptoms of depression over the past two weeks. The higher the total score, the more severe the depression.
Beck Depression Inventory (BDI-II) | 14 months after baseline (follow-up)
  The Beck Depression Inventory (BDI-II) is the 1996 revision of the BDI created by Dr. Aaron T. Beck, which is one of the most widely used self-report questionnaires measuring the severity of depression. The 21 multiple-choice items address the severity of 21 typical symptoms of depression over the past two weeks. The higher the total score, the more severe the depression.
Quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | 4 months after baseline
  The WHOQOL-BREF self-report questionnaire is the abbreviated 26-item version of the WHOQOL-100. It assesses the perceived quality of life (e.g. "To what extent do you feel your life to be meaningful?"). Quality of life is defined by the WHO as "…individuals' perceptions of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns."
Quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | 8 months after baseline
  The WHOQOL-BREF self-report questionnaire is the abbreviated 26-item version of the WHOQOL-100. It assesses the perceived quality of life (e.g. "To what extent do you feel your life to be meaningful?"). Quality of life is defined by the WHO as "…individuals' perceptions of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns."
Quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | 14 months after baseline (follow-up)
  The WHOQOL-BREF self-report questionnaire is the abbreviated 26-item version of the WHOQOL-100. It assesses the perceived quality of life (e.g. "To what extent do you feel your life to be meaningful?"). Quality of life is defined by the WHO as "…individuals' perceptions of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns."
Perceived Stress Questionnaire (PSQ20) | 4 months after baseline
  The Perceived Stress Questionnaire (PSQ20) is the abbreviated 20-item version of the PSQ (Levenstein et al., 1993) and assesses self-reported experienced stress.
Perceived Stress Questionnaire (PSQ20) | 8 months after baseline
  The Perceived Stress Questionnaire (PSQ20) is the abbreviated 20-item version of the PSQ (Levenstein et al., 1993) and assesses self-reported experienced stress.
Perceived Stress Questionnaire (PSQ20) | 14 months after baseline (follow-up)
  The Perceived Stress Questionnaire (PSQ20) is the abbreviated 20-item version of the PSQ (Levenstein et al., 1993) and assesses self-reported experienced stress.

CONTACTS AND LOCATIONS:
Overall Officials: Hansjoerg Znoj, Prof. Dr. phil., Study Chair — Dep. of Clinical Psychology and Psychotherapy, University of Berne; Helene Hofer, Dr. phil., Study Director — Bern University Hospital, Outpatient Clinic for Cognitive and Restorative Neurology; Martin Grosse Holtforth, Prof. Dr. phil., Study Director — University of Zurich, Dep. of Psychology, Research Unit Psychotherapy for Depression; Rene M Mueri, Prof. Dr. med., Study Director — Bern University Hospital, Outpatient Clinic for Cognitive and Restorative Neurology; Eveline Frischknecht, lic. phil., Principal Investigator — Dep. of Clinical Psychology and Psychotherapy, University of Berne
Locations (1):
- Dep. of clinical psychology and psychotherapy, University of Berne, Bern, Switzerland

REFERENCES:
- See also: Related Info — http://oscar.online-therapy.ch